CLINICAL TRIAL: NCT02407015
Title: A Randomised Control Trial to Evaluate the Effect of 3D Autostereoscopic Video-game Play on the Total Horizontal Fusional Vergence Amplitudes of 7 to 11 Year Old Children
Brief Title: The Effect of 3D Autostereoscopic Video-game Play on the Visual Fatigue in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Responsible Party: Principal Investigator, Mrs Louisa Haine, Lead Orthoptic Clinical Tutor, University of Sheffield
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: URMS 138673
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Visual Fatigue
MeSH Terms: conditions — Asthenopia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3D gameplay (Active Comparator): Participants will play a game for 30 minutes on the Nintendo 3DS in 3D.
  Interventions: Other: Nintendo 3DS gameplay
- 2D gameplay (Active Comparator): Participants will play a game for 30 minutes on the nintendo 3DS in 2D.
  Interventions: Other: Nintendo 3DS gameplay

INTERVENTIONS:
Other: Nintendo 3DS gameplay

SUMMARY:
This study aims to examine the specific effect that 3D game play has on the control of the eyes horizontal movements. It will examine the youngest group of consumers this technology is marketed to, 7 to 11-year-olds and no children under 7 years of age will be recruited to this study as per Nintendo's hardware guidelines, which recommends that children under 7 years of age not play in 3D mode. It will examine the effect of playing in 3D for 30 minutes on horizontal fusional amplitudes compared with a control group playing in 2D for 30 minutes.

DETAILED DESCRIPTION:
This study will be a prospective blind randomised control trial. The participants will be randomised into one study group, with participants playing a game in 3D; and a control group, with participants playing the same game in 2D. The study is blind due to the use of an independent assessor, reducing testing bias by ensuring that the tester does not know the randomisation results. The known dependant variables are the total horizontal fusional amplitudes at 1/3m and 6m and the independent variable is the use of 2D or 3D game play.

ELIGIBILITY:
Inclusion Criteria:

* Male and female 7 to 11-year-olds with no prior history of binocular vision / ocular motility dysfunction.

Exclusion Criteria:

* Corrected visual acuity of less than 0.000 tested with SLT at 3m.

  * Interocular visual acuity difference of 0.100 (tested with SLT) or greater, which could indicate the presence of Amblyopia.
  * The presence of any manifest deviation (Tropia).
  * Presence of any ocular motility dysfunction, which affects primary position.
  * Reduced binocular convergence of 10 centimetres or less.
  * Stereoacuity of less than 170" (this may indicate the presence of a microtropia or other undiagnosed pathology).
  * Any prior or existing medical history of epilepsy or seizures.
  * Any prior or existing medical history of repetitive strain injury.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2014-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in horizontal fusional amplitude | Immediately following gameplay

CONTACTS AND LOCATIONS:
Overall Officials: Louisa A Haine, BSc, Principal Investigator — University of Sheffield
Locations (1):
- Cambridge University Hospitals NHS trust, Cambridge, Cambridgeshire, United Kingdom